CLINICAL TRIAL: NCT06538597
Title: Online Mindful Self-Compassion Training for Medical Students: an Exploratory Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Simpson (Other)
Responsible Party: Sponsor-Investigator, Robert Simpson, Assistant Professor, Department of Medicine, University of Toronto
Organization: University of Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 00046332
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-08

CONDITIONS: Self-Compassion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self-compassion intervention (Experimental): 6-week manualized online Self-Compassion for Healthcare Communities course
  Interventions: Behavioral: Self-compassion intervention (Self-Compassion for Healthcare Communities course)

INTERVENTIONS:
Behavioral: Self-compassion intervention (Self-Compassion for Healthcare Communities course) — An online 6-week mindful self-compassion course with weekly sessions.

SUMMARY:
The goal of this clinical trial is to develop and investigate a compassion-based intervention (Self-Compassion for Healthcare Communities (SCHC) course) in medical students. The main objectives are:

1. Explore the feasibility of trial processes including recruitment, adherence, retention, and follow-up
2. Explore the experiences of medical students with the Compassion-based intervention, including perceived effects, barriers and facilitators to participation, suggestions for improvement
3. Determine potential effects on burnout, compassion fatigue, compassion satisfaction, self-compassion, compassion for others, empathy, mindfulness, perceived stress, and emotional regulation.

Participants will be asked to take part in a 6-week online Self-Compassion for Healthcare Communities course and report changes in levels of burnout, compassion fatigue, compassion satisfaction, self-compassion, compassion for others, empathy, mindfulness, perceived stress, and emotional regulation from pre- to post-intervention and at 3-month follow-up. Additionally, participants will be asked to take part in a semi-structured interview to explore their experiences with the course, perceived effects, and suggestions for improvement.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in first or second-year of the MD or MD/PhD program at the University of Toronto,
2. Over 18 years of age,
3. Able to speak, read, and write in English,
4. Willing to take part in the SCHC course for up to the full 6-week duration,
5. Willing to complete all study related questionnaires

Exclusion Criteria:

1. Those already having completed a mindful self-compassion course or Mindfulness based-intervention (Mindfulness-based stress reduction or Mindfulness-based cognitive therapy) within the past 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 4 months
  The investigators will measure the number of participants eligible for and recruited to the study.
Retention | 4 months
  The investigators will measure the percentage of participants who complete outcome data.
Adherence | 4 months
  The investigators will measure the number of participants who completed the Self-Compassion for Healthcare Communities course.
Follow-up rates | 4 months
  The investigators will measure the percentage of participants who complete outcome measures pre-intervention, post-intervention, and at 3 months post-intervention.

SECONDARY OUTCOMES:
Professional Quality of Life Scale (ProQOL) Version 5 | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures the positive and negative effects of one's compassion for those that they help. Includes with subscales for compassion satisfaction and compassion fatigue (including burnout). Answers are assessed using a 5-point Likert scale, with higher scores on the compassion satisfaction sub-scale indicating higher compassion satisfaction, and higher scores on compassion fatigue sub-scale indicating higher burnout.
Self-Compassion Scale - Short Form | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures how one typically acts towards themselves in difficult times. The total score ranges from a 1-5, with higher scores representing high self-compassion.
Relational Compassion Scale | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measure's ones tendencies for receiving and providing relational compassion. Answers are assessed using a 4-point Likert scale. Higher scores represent higher compassion for self and others.
The Brief Interpersonal Reactivity Index | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures the different ways that people may think about their lives. Answers are assessed using a 5-point Likert scale, with higher scores representing higher empathic responsiveness.
Five Facet Mindfulness Questionnaire: Short Form | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures one's tendencies to engage in mindfulness practices. Answers are assessed using a 5-point Likert scale, with higher scores representing more mindfulness.
Perceived Stress Scale-10 | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures one's thoughts and feelings pertaining to stress. The total score can range from 0-40, with higher scores indicating higher perceived stress.
Difficulties in Emotion Regulation Scale - Short Form | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures emotion regulation. Answers are assessed using a 5-point Likert scale. Higher values indicate greater difficulties in emotion regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Simpson, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No